CLINICAL TRIAL: NCT05491551
Title: Brief Training for Heavy Drinking Young Adults: Regulation of Alcohol Craving
Brief Title: Alcohol-ROC-Training
Acronym: A-ROC-T
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2000029394; 1R01AA029137-01 (NIH)
Record Dates: First submitted 2022-07-07; First posted 2022-08-08 (Actual); Last update posted 2025-04-11 (Actual); Status verified 2025-04

CONDITIONS: Binge Drinking; Heavy Drinking; Young Adult; Heavy Drinker
Keywords: Binge Drinking; Heavy Drinking; Young Adult; Heavy Drinker; Regulation of Craving; Cognitive Behavioral Therapy; Neurocognitive Training; Mindfulness-Based Therapy
MeSH Terms: conditions — Binge Drinking; Alcoholic Intoxication

STUDY DESIGN:
Intervention Model Description: Randomized Control Trial
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Mindfulness-Based Treatment (Experimental): Using mindfulness and meditative strategies to control craving
  Interventions: Behavioral: Mindfulness-Based Treatment-Regulation of Craving
- Cognitive Behavioral Therapy (Experimental): Thinking of negative consequences to control craving
  Interventions: Behavioral: Cognitive-Based Therapy-Regulation of Craving
- Control (No Intervention): No regulatory strategy

INTERVENTIONS:
Behavioral: Mindfulness-Based Treatment-Regulation of Craving — Participants will be trained in using the MBT-based mindfulness strategy as described above ("notice craving and accept the feeling without judgment or reaction"). Participants will then be instructed to think of accepting and non-reactive responses when they see the instruction "ACCEPT" during ROC-T. On each trial, participants will receive an instruction and then be exposed to a novel alcohol image for 6 seconds. On 25% of the trials, they will see the LOOK instruction, and be allowed to experience craving (as baseline). On 75% of the trials, participants will see ACCEPT and then practice thinking about the negative consequences of drinking. After the picture disappears, they will rate their craving on every trial using a 1-5 Likert scale.
  Other Names: MBT-ROC
  Arms: Mindfulness-Based Treatment
Behavioral: Cognitive-Based Therapy-Regulation of Craving — Participants will be trained in using the CBT strategy by first considering and reading about the negative consequences of drinking. Participants will then be instructed to think of those negative consequences ("Focus on the negative consequences associated with drinking)" when they see the instruction "REFRAME" during ROC-T.On each trial, participants will receive an instruction and then be exposed to a novel alcohol image for 6 seconds. On 25% of the trials, they will see the LOOK instruction, and be allowed to experience craving (as baseline). On 75% of the trials, participants will see REFRAME and then practice thinking about the negative consequences of drinking. After the picture disappears, they will rate their craving on every trial using a 1-5 Likert scale
  Other Names: CBT-ROC
  Arms: Cognitive Behavioral Therapy

SUMMARY:
The goal of the proposed study is to examine whether brief training in regulation of craving (ROC-T) affects alcohol drinking. The study will consist of a basic screening (phone and online), and in person visit to determine eligibility and conduct pre-intervention baseline assessments, 1-4 training (ROC-T) visits, a post-intervention assessment visit, and 1-2 phone/online follow up assessments.The two active conditions of ROC-T are based on cognitive-behavioral treatments (CBT) and mindfulness-based treatments (MBT).

DETAILED DESCRIPTION:
This is a Stage 1B Randomized-Controlled Trial (RCT). 177 heavy drinking young adult participants will be randomized to 4 x 45-minute web-based sessions of (1) CBT-ROC-T training, (2) MBT-ROC-T, or (3) CONTROL (no strategy) delivered over three weeks. Participants will be enrolled for 16 weeks (three weeks pre-, three weeks during, and ten weeks post-intervention).

ELIGIBILITY:
Inclusion Criteria:

(1) Young adults ages 18-26 years, who (2) report ≥ 3 heavy drinking days (i.e., heavy drinking defined by >3 drinks for women, >4 drinks for men) in the prior month; (3) are motivated to quit or reduce drinking; (4) are fluent in English and have a 6th grade or higher reading level; (5) have access to a computer with working internet; (6) use a working smartphone; (7) can commit to the full length of the protocol; and (8) are willing to be randomized to intervention condition.

Exclusion Criteria:

(1) Current (past 12 months) clinically-severe alcohol use disorder (AUD; e.g., history of seizures, delirium, or hallucinations during withdrawal) or current severe alcohol withdrawal; (2) Current (past 12 months) clinically-severe substance use disorder (except tobacco) or current severe drug withdrawal; (3) serious other psychiatric illness by history or examination; (4) severe or unstable physical disease within the past 6 months; (5) psychoactive medications (e.g., mood stabilizers) that have not been at a stable dose unless determined to be on a stable dose of medication by the study psychiatrist; (6) current use of any investigational medication; (7) color blindness; (8) biological females who are pregnant; and (9) notable dislike to any particular type of alcoholic beverage depicted in study stimuli; (10) Participants who will not complete at least 70% of past day EMA reports in the pre-intervention phase will not be randomized; (11) Participants who cannot understand or follow study-related instructions (e.g., unable to correctly use the intervention strategies, indicate lack of understanding of study instructions despite multiple attempts).

Ages: 18 Years to 26 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 177 (Estimated)
Dates: Start 2022-09-28 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Change in frequency of heavy drinking days | From baseline to 2-weeks post-intervention and to the 10-week follow-up
  Self-reports of daily alcohol use via smartphone-based ecological momentary assessment (EMA) is the primary source for this outcome variable, with Timeline Follow-Back (TLFB) data inserted to replace missing data from EMA. A heavy drinking day is defined as more than 3 or 4 standard drinks per day for women/men.
Change in average estimated blood alcohol concentration (eBAC) per drinking day | From baseline to 2-weeks post-intervention and to the 10-week follow-up
  Daily self-reports of alcohol use via smartphone-based ecological momentary assessment (EMA) is the primary source for this outcome variable, with Timeline Follow-Back (TLFB) data inserted to replace missing data from EMA. Estimated blood alcohol concentration (eBAC) is based on number of standard drinks reported per day, duration of drinking, and total body water (based on sex, age, height, and weight).

SECONDARY OUTCOMES:
Change in alcohol-related negative consequences | From baseline to 2-weeks post-intervention and the 10-week follow-up
  Daily self-reports of alcohol-related negative consequences (Brief Young Adult Alcohol Consequences Questionnaire) via smartphone-based ecological momentary assessment (EMA) is the primary source for this outcome variable. Total scores range from 0 to 24, with higher scores indicating greater alcohol-related negative consequences.
Reduction in World Health Organization (WHO) drinking risk level | From baseline to 2-weeks post-intervention and the 10-week follow-up
  Drinking risk levels are based on grams of pure alcohol per day in a given period and include abstinent (0 grams males/females), low risk (1 to 40g males/1 to 20g females), medium risk (41 to 60g males/21 to 40g females), high risk (61 to 100g males/41 to 60g females), or very high risk (greater to or equal to 101g males/61g females).

OTHER OUTCOMES:
Change in momentary alcohol craving in daily life | From baseline to 2-weeks post-intervention and the 10-week follow-up
  Twice daily self-reports of momentary craving for alcohol via smartphone-based ecological momentary assessment (EMA). Alcohol craving scores range from 0 to 10, with higher scores indicating greater alcohol craving.
Change in momentary acceptance of craving in daily life | From baseline to 2-weeks post-intervention and the 10-week follow-up
  Twice daily self-reports of momentary acceptance of alcohol craving via smartphone-based ecological momentary assessment (EMA). Acceptance of alcohol craving scores range from 0 to 10, with higher scores indicating greater acceptance of alcohol craving.
Change in momentary reframing of craving in daily life | From baseline to 2-weeks post-intervention and the 10-week follow-up
  Twice daily self-reports of momentary reframing of alcohol craving via smartphone-based ecological momentary assessment (EMA). Reframing of alcohol craving scores range from 0 to 10, with higher scores indicating greater reframing of alcohol craving.
Change in momentary craving during Regulation of Craving (ROC) task | From baseline ROC task to post-intervention ROC task (approximately 3 weeks)
  The ROC task involves viewing a series of alcohol images and following various instructions on particular trial when an alcohol image is shown. Participants report self-reported craving after each trial. There are 3 types of trials: 1) LOOK = look at alcohol image, 2) ACCEPT = use acceptance strategy, and 3) REFRAME = use the reframing strategy.

CONTACTS AND LOCATIONS:
Overall Officials: Hedy Kober, Ph.D., Principal Investigator — Yale University
Locations (1):
- Yale University, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: Yes
We will adhere to the NIH Grants Policy on Sharing of Unique Research Resources.
  In compliance with HIPAA and Yale Human Investigation Committee standards, any data sets that will be shared will not include any personally identifiable information. Requests for data sharing will be considered within the context of ongoing and planned research being performed within the research group at Yale in order to avoid duplication of effort and overlap in data analysis that might compromise communication of findings. Data to be shared will be de-identified and transmission electronically and securely, as we have done previously with investigators at other institutions.